CLINICAL TRIAL: NCT03147781
Title: The Effect of Auricular Therapy on Lactation: A Pilot Study
Brief Title: Auricular Therapy for Postpartum Lactation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSEARS20170214003
Record Dates: First submitted 2017-04-27; First posted 2017-05-10 (Actual); Last update posted 2018-06-12 (Actual); Status verified 2018-06

CONDITIONS: Lactation; Cesarean
Keywords: auriculotherapy, human milk, breastfeeding, lactogenesis
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard care (No Intervention): Participants in this group only receive standard post-cesarean care of the study hospital. It includes mobility restraint, foley retention, IV fluid infusion, oral intake instructions, oral pain medications routine, and breastfeeding practice.
- Sham AT with Medulla Junci (Sham Comparator): Participants in this group receive auricular tape with Medulla Junci in addition to standard post-cesarean care during the early 96 postpartum hours.
  Interventions: Device: Sham AT with Medulla Junci
- True AT with magnetic pellets (Experimental): Participants in this group receive auricular tape with magnetic pellets in addition to standard post-cesarean care during the early 96 postpartum hours.
  Interventions: Device: True AT with magnetic pellets

INTERVENTIONS:
Device: True AT with magnetic pellets — Magnetic pellets are affixed onto pre-selected auricular acupoints with tape.The treatment was initiated within 4 to 8 hours post cesarean for 96 hours during the hospital stay.
  Arms: True AT with magnetic pellets
Device: Sham AT with Medulla Junci — Medulla Junci segments are crumbled into ball-shape and then attached to the pre-selected auricular acupoints with tape. The treatment was initiated within 4 to 8 hours post cesarean for 96 hours during the hospital stay.
  Arms: Sham AT with Medulla Junci

SUMMARY:
The aim of this study is to function as a pilot study in evaluating the effects of auricular therapy (AT) on lactation for women in the immediate post cesarean period while examining the feasibility of the three-parallel-arm, sham-controlled randomized design. The study hypothesizes that post cesarean women who receive AT with standard care for 96 hours postpartum have earlier onset of lactogenesis II and larger milk production when compared with women who receive sham AT with standard care or standard care alone.

DETAILED DESCRIPTION:
Breastfeeding has been of major concern in maternal-child healthcare. Challenges posed by cesarean delivery can have negative impacts on breastfeeding. Efforts to facilitate, support, and sustain breastfeeding have been investigated to a great extent by researchers from a variety of disciplines. In the field of Traditional Chinese Medicine (TCM), a number of clinical studies have been carried out to study the effect of auricular therapy (AT) on postpartum lactation over the years. Limitations in the evidence that currently exists include the lack of randomization, sham-controlled treatment, blinding and/or no valid outcome measures. Given that such information is important for maternal-child health and clinical practice, the study has set out to conduct a pilot trial which employs randomized, single-blinded, and sham group design that examines relevant outcomes using valid measurement.

A total of 96 post cesarean participants have been randomly assigned to one of three treatment conditions: (1) standard care (n=32); (2) standard care with Medulla Junci adhesive on auricular acupoints (n=32); (3) standard care with magnetic pellets adhesive on auricular acupoints (n=32). The standard care group participants only received the standard post cesarean care of the study hospital without any additional therapies. The same set of six pre-specified auricular points were adopted for both Medulla Junci and magnetic pellets groups. The treatment was initiated within 4 to 8 hours post cesarean for 96 hours during their hospital stay at a maternal hospital in Kaohsiung, Taiwan.

Milk production and onset of lactogenesis II have been used as primary outcome variables for the evaluation of the effectiveness of AT. Milk production is determined by the summed value of infant test weighing measurements and expressed breast milk. Maternal perceptions of breast fullness, swelling, leakage, or tingling are the indicator of onset of lactogenesis II. The secondary outcome measures are infant behaviors of observed swallowing and rooting during breastfeeding, neonatal weight gain, and frequencies of urination and defecation of the infant.

Numeric rating scales have been used to measure the effect of the possible mediating variables, i.e., pain and stress. Potential confounding variables have been controlled by either stratified randomization and exclusion criteria or monitored during the study period. Treatment expectation and satisfaction toward AT have been assessed in order to examine their relationship with therapy outcomes. Main components of study feasibility, i.e., recruitment, retention, and acceptance, have been evaluated. Participants also have been contacted to acquire their one and three-month breastfeeding practice status.

ELIGIBILITY:
Inclusion Criteria:

1. Mothers and their term (37-42 weeks) and singleton infants
2. Has cesarean section at the study hospital, irrespective of the reason for cesarean (primary, repeated, indicated, elective, scheduled, unscheduled, emergency, or non-emergency)
3. Intent to stay hospitalized for at least 96 hours after birth
4. Intent to breastfeed
5. Able to communicate with Chinese, Taiwanese, or English

Exclusion Criteria:

1. Mothers and their preterm infants (<37 weeks), postterm infants (>42weeks)
2. Infants who are not able to be breastfed
3. Acute and chronic maternal health problems that can affect lactation. 3.1 Acute illness and infections: e.g. tuberculosis, Group B Streptococcus, Methicillin-Resistant Staphylococcus Aureus (MRSA), etc. 3.2 Alternations in endocrine and metabolic functioning: hypothyroidism, hypopituitarism, diabetes, Sheenhan's syndrome, gestational ovarian theca lutein cysts, polycystic ovarian syndrome. 3.3 Breast-related problems, e.g., breast surgery, injury, and cancer, etc. 3.4 Perinatal conditions: placental retention, dysfunctional uterine bleeding.
4. Skin conditions in the ear such as rashes, moles, scars, irritation or ear abrasions.
5. Has an implanted electrical device (for example, a pacemaker).
6. Has earrings on the selected auricular acupoints.
7. Had been receiving auricular therapy within the past six months.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2017-04-07 (Actual); Primary Completion 2018-03-08 (Actual); Study Completion 2018-06-08 (Actual)

PRIMARY OUTCOMES:
Onset of lactogenesis II | up to five postpartum days
  Maternal perception of breast symptoms of lactation, i.e., breast fullness, swelling, leakage, or tingling, are employed in identifying onset of lactogenesis II. Assessment of maternal perception began within 4 to 8 hours postpartum. Participants was instructed to record the approximate time when breast symptoms of lactation first noticed. They was interviewed regarding these breast symptoms twice daily during their hospital stay.
Change of Milk production | first five postpartum days
  Milk production is determined by the summed value of infant test weighing measurements and expressed breast milk. Test weighing procedure, whereby the infant is weighted under exactly the same clothing and diaper immediately before and after feeding to estimate milk intake during breastfeeding.

SECONDARY OUTCOMES:
Neonatal behaviors of swallowing and rooting during breastfeeding. | first five postpartum days
  Infants were observed by the study assessor during breastfeeding once daily. The result obtained from this outcome will assist the evaluation of milk production change.
Neonatal weight | first five postpartum days
  The data were collected from the nursery record.The result obtained from this outcome will assist the evaluation of milk production change.
Frequencies of urination and defecation | first five postpartum days
  The data were collected from the nursery record.The result obtained from this outcome will assist the evaluation of milk production change.

CONTACTS AND LOCATIONS:
Overall Officials: Lorna KP Suen, Ph.D, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- Love Saint Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No